CLINICAL TRIAL: NCT01506453
Title: Therapeutic Interventions For Peripheral Neuropathy/Neuropathic Pain Induced By Vincristine Treatment For Childhood Acute Lymphoblastic Leukemia (ALL) On Total XVI Protocol
Brief Title: Therapeutic Interventions For Pain Induced By Vincristine Treatment For Childhood Acute Lymphoblastic Leukemia (ALL)
Acronym: TINALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TINALL; NCI-2012-00413 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2012-01-04; First posted 2012-01-10 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-04

CONDITIONS: Acute Lymphoblastic Leukemia; Neuropathy; Neuropathic Pain
Keywords: Acute Lymphoblastic Leukemia; Neuropathy; Neuropathic Pain; Vincristine; TOTAL XVI Protocol
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neuralgia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Active Comparator): Active treatment arm.
  Interventions: Drug: gabapentin
- Placebo (Placebo Comparator): Placebo arm.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: gabapentin — Participants randomized to the active treatment arm will receive gabapentin 20mg/kg/day PO divided into 3 doses and rounded to the nearest 100 mg for capsules and 10 mg for liquid preparation.
  Other Names: Treatment Arm
  Arms: Gabapentin
Drug: placebo — Participants randomized to the placebo treatment arm will receive look-alike capsules or liquid in a respective capsule size or liquid measure equivalent to the active treatment arm, but which contain no active treatment.
  Other Names: Placebo Arm
  Arms: Placebo

SUMMARY:
Neuropathic pain / peripheral neuropathy (NP/PN) is a known painful complication of vincristine (VCR) therapy; evidence supporting the best treatment plan for pediatric patients is limited. Gabapentin is frequently used for VCR-related NP/PN, with variable dosing and scheduling regimens, and with varying measures of success. The hypothesis of the study is that gabapentin will reduce the severity of NP/PN in patients receiving vincristine during treatment for ALL on the Total XVI protocol (or for those being treated "as per TOTXVI protocol"), as measured by two outcome measures: the daily dose of morphine used as needed for pain in addition to either gabapentin or placebo, as randomized, and the pain scores assessed daily.

DETAILED DESCRIPTION:
Patients with ALL on Total XVI ((or for those being treated "as per TOTXVI protocol") who experience NP/PN after specific doses of vincristine are eligible to enroll in the study as soon as the diagnosis of NP/PN related to VCR is established. The qualifying doses of vincristine have been selected because they fall in the schedule of weekly vincristine doses as per Total XVI, and 2 additional weekly vincristine doses are anticipated according to the protocol. Participants will be randomized to receive gabapentin or placebo upon enrollment. Morphine will be available to both groups as needed for pain at any time on the study. At the time of enrollment, and daily thereafter until completion of the study drug, data will be collected for pain assessment, and the daily dose of oral morphine used will be collected. Data regarding the pain type, quality, and location, as well as treatments used to manage pain will be assessed on a daily basis for the diagnostic event and for the period following the next two administrations of VCR treated with the study drug.

Primary Objective: To assess the analgesic efficacy of gabapentin in controlling VCR-related NP/PN in participants with ALL, by comparing the morphine daily dose (mg/kg/day) used to control NP/PN as a primary or a rescue regimen in the gabapentin vs. placebo groups.

Secondary Objective: To compare the pain scores in the gabapentin and placebo groups as recorded by pain score right now and pain score average for previous 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Participant is enrolled on Total XVI or who are being treated "as per TOTXVI protocol"
* Participant is 1 year of age or older
* Participant has symptoms of NP/PN with onset no more than 7 days after one of the following vincristine doses ± 3 days: protocol week 1, week 2 (induction), week 7 (reinduction I), or week 17 (reinduction II).
* Patient is expected to receive 2 doses of vincristine in weekly intervals as outlined by the Total XVI protocol (or for those being treated "as per TOTXVI" protocol) while on study drug (i.e. no known dosage reductions or planned missed doses).

Participant is able and willing to take oral medications.

Exclusion Criteria:

* Previous participation in this study
* Participant is receiving gabapentin for another indication at the time of diagnosis of NP/PN or has received gabapentin previously.
* Pregnancy. Female participants of childbearing potential must have documented negative urine or serum pregnancy test result not older than 7 days. Male patients with reproductive potential will be counseled not to procreate during the study.
* Impaired renal function: decreased eGFR (<60ml/min/1.73m^2 as estimated by the revised Schwartz equation)
* Participant has allergy or other contraindication for either morphine or gabapentin therapy.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doralina Anghelescu, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 participants were enrolled and screened between January 2012 and October 2016.
Pre-assignment Details: The remaining 51 participants were randomized to take gabapentin or placebo.
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 25 | 26
Completed | 25 | 24
Not Completed | 0 | 2
Not completed — Withdrawal prior to treatment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.88 (5.69) | 7.08 (3.90) | 7.48 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 14 | 16 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Baseline Measures: Asian and White | 0 | 1 | 1
  Baseline Measures: Black | 1 | 2 | 3
  Baseline Measures: Black and White | 1 | 2 | 3
  Baseline Measures: White | 23 | 21 | 44
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 26 | 51
Daily "pain score right now" [Mean (Standard Deviation); unit: units on a scale] — Pre-treatment (baseline) and (pain score right now) will be obtained. The scores are used in stratified randomization. Infants and toddlers (less than age 4 years) or other children who cannot self report, use the FLACC Scale . Self report using a numeric scale 0-10 without reference to Faces Pain Scale-Revised (FPS-R) Pain score 0 means no pain and 10 means worst pain. The scale information for the FLACC and FPS-R scales are similar. Population: 2 of 26 patients in the placebo group did not receive the placebo and therefore no data was generated based on them.
  units on a scale
    number analyzed (Participants) | 25 | 24 | 49
    (all) | 3.12 (1.86) | 3.58 (1.42) | 3.35 (1.65)
baseline pain score last 24 hours [Mean (Standard Deviation); unit: units on a scale] — Pre-treatment (baseline) and (pain score right now) will be obtained. The scores are used in stratified randomization. Infants and toddlers (less than age 4 years) or other children who cannot self report, use the FLACC Scale . Self report using a numeric scale 0-10 without reference to Faces Pain Scale-Revised (FPS-R) Pain score 0 means no pain and 10 means worst pain. The scale information for the FLACC and FPS-R scales are similar. Population: 2 of 26 patients in the placebo group did not receive the placebo and therefore no data was generated based on them.
  units on a scale
    number analyzed (Participants) | 25 | 24 | 49
    (all) | 4.08 (1.66) | 4.31 (1.76) | 4.20 (1.70)

OUTCOME MEASURES:

1. Primary Outcome: Daily Total Dose of Oral Morphine (mg/kg/Day).
Description: The response to therapy will be measured by pain intensity scores and daily use of morphine doses for breakthrough pain as described in the study objectives. Daily assessments will continue during treatment with the study drug (gabapentin or placebo) irrespective of patient response to study treatment. and toddlers (less than age 4 years) or other children who cannot self report, use the FLACC Scale Score each component as a subscore (face, legs, activity, cry, consolability) Total subscores to determine FLACC score Older children (ages 4 to 7 years) who can self-report, use the Faces Pain Scale-Revised (FPS-R) Ages >7 years, Self report using a numeric scale 0-10 without reference to Faces Pain Scale-Revised (FPS-R) Pain score 0 means no pain and 10 means worst pain. The scale information for the FLACC and FPS-R scales are similar.
Time Frame: Daily beginning day 1 for a maximum of 21 days.
Population: The daily morphine dosage will be modeled as longitudinal observations with treatment (gabapentin vs. placebo) group, and if necessary, other clinical factors such as age category for pain assessment (0-3yr, 4-7yr, >7yr), baseline pain score, and ALL risk classification, as explanatory factors, using repeated measure linear models
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 24
mg/kg/day
  Day 1: number analyzed (Participants) | 9 | 6
  Day 1 | 0.38267 (0.28921) | 0.27433 (0.19299)
  Day 2: number analyzed (Participants) | 13 | 16
  Day 2 | 0.43685 (0.33788) | 0.31816 (0.16012)
  Day 3: number analyzed (Participants) | 15 | 16
  Day 3 | 0.37281 (0.32935) | 0.27961 (0.18509)
  Day 4: number analyzed (Participants) | 14 | 12
  Day 4 | 0.40384 (0.32469) | 0.35343 (0.18688)
  Day 5: number analyzed (Participants) | 13 | 9
  Day 5 | 0.37662 (0.31263) | 0.37920 (0.22471)
  Day 6: number analyzed (Participants) | 14 | 9
  Day 6 | 0.45679 (0.45450) | 0.43972 (0.19838)
  Day 7: number analyzed (Participants) | 14 | 11
  Day 7 | 0.50961 (0.43643) | 0.37181 (0.22883)
  Day 8: number analyzed (Participants) | 15 | 10
  Day 8 | 0.50767 (0.53570) | 0.38188 (0.28251)
  Day 9: number analyzed (Participants) | 16 | 10
  Day 9 | 0.49234 (0.33366) | 0.34524 (0.20164)
  Day 10: number analyzed (Participants) | 13 | 10
  Day 10 | 0.44392 (0.37244) | 0.34660 (0.15843)
  Day 11: number analyzed (Participants) | 15 | 9
  Day 11 | 0.50981 (0.67516) | 0.29937 (0.14111)
  Day 12: number analyzed (Participants) | 13 | 11
  Day 12 | 0.57798 (0.51346) | 0.40090 (0.21956)
  Day 13: number analyzed (Participants) | 14 | 9
  Day 13 | 0.68183 (0.51698) | 0.45933 (0.32854)
  Day 14: number analyzed (Participants) | 16 | 9
  Day 14 | 0.53028 (0.57870) | 0.34957 (0.15460)
  Day 15: number analyzed (Participants) | 15 | 11
  Day 15 | 0.55939 (0.69755) | 0.36731 (0.23170)
  Day 16: number analyzed (Participants) | 11 | 5
  Day 16 | 0.37643 (0.37817) | 0.48481 (0.37075)
  Day 17: number analyzed (Participants) | 7 | 3
  Day 17 | 0.38837 (0.30190) | 0.54960 (0.47579)
  Day 18: number analyzed (Participants) | 4 | 1
  Day 18 | 0.65013 (0.96603) | 0.13605 (NA) — Measure of dispersion not calculated.
  Day 19: number analyzed (Participants) | 3 | 3
  Day 19 | 0.84586 (1.08656) | 0.14123 (0.00740)
  Day 20: number analyzed (Participants) | 2 | 1
  Day 20 | 1.12358 (1.37790) | 0.15108 (NA) — Measure of dispersion not calculated.
  Day 21: number analyzed (Participants) | 1 | 0
  Day 21 | 0.14981 (NA) — Measure of dispersion not calculated. |

2. Secondary Outcome: Pain Scores Right Now
Description: A score ranging from 0 to 10, measured by age appropriate validated pain scale. Because there was only one patient during day 21 time point for this treatment group, the mean and standard deviation could not be calculated. Infants and toddlers (less than age 4 years) or other children who cannot self report, use the FLACC Scale Score each component as a subscore (face, legs, activity, cry, consolability) Total subscores to determine FLACC score Older children (ages 4 to 7 years) who can self-report, use the Faces Pain Scale-Revised (FPS-R) Ages >7 years, Self report using a numeric scale 0-10 without reference to Faces Pain Scale-Revised (FPS-R) Pain score 0 means no pain and 10 means worst pain.The scale information for the FLACC and FPS-R scales are similar.
Time Frame: Daily beginning day 1 through a maximum of 21 days.
Population: There were participants in the Gabapentin and Placebo groups that did not have pain assessments at various time points. Pain score was 0 for each placebo participant on days 19, 20 and 21.
Measure: Mean (Standard Deviation); unit: score on a scale 0-10
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 24
score on a scale 0-10
  Day 1: number analyzed (Participants) | 25 | 23
  Day 1 | 1.64000 (1.89033) | 1.69565 (2.09837)
  Day 2 | 2.00000 (2.19848) | 1.16667 (1.57885)
  Day 3 | 1.88000 (2.60320) | 0.75000 (1.25974)
  Day 4 | 1.92000 (2.64449) | 0.83333 (1.30773)
  Day 5 | 1.64000 (1.97653) | 1.00000 (1.44463)
  Day 6 | 1.40000 (1.75594) | 0.79167 (1.38247)
  Day 7 | 2.20000 (2.17945) | 0.91667 (1.50121)
  Day 8: number analyzed (Participants) | 25 | 23
  Day 8 | 1.32000 (1.90875) | 0.56522 (1.23679)
  Day 9: number analyzed (Participants) | 25 | 23
  Day 9 | 1.48000 (2.06398) | 0.86957 (1.63219)
  Day 10: number analyzed (Participants) | 25 | 23
  Day 10 | 1.16000 (1.65025) | 0.39130 (0.83878)
  Day 11: number analyzed (Participants) | 25 | 23
  Day 11 | 1.16000 (1.90788) | 0.82609 (1.26678)
  Day 12: number analyzed (Participants) | 23 | 23
  Day 12 | 1.21739 (1.88189) | 1.00000 (1.50756)
  Day 13: number analyzed (Participants) | 23 | 23
  Day 13 | 1.04348 (1.46095) | 0.69565 (1.39593)
  Day 14: number analyzed (Participants) | 23 | 23
  Day 14 | 0.82609 (1.11405) | 0.52174 (1.23838)
  Day 15: number analyzed (Participants) | 22 | 23
  Day 15 | 0.90909 (1.63034) | 0.60870 (1.23359)
  Day 16: number analyzed (Participants) | 17 | 16
  Day 16 | 1.29412 (1.99263) | 0.31250 (0.87321)
  Day 17: number analyzed (Participants) | 15 | 14
  Day 17 | 0.40000 (0.91026) | 0.21429 (0.80178)
  Day 18: number analyzed (Participants) | 11 | 12
  Day 18 | 1.45455 (2.54416) | 0.25000 (0.86603)
  Day 19: number analyzed (Participants) | 5 | 5
  Day 19 | 1.00000 (1.41421) | 0 (0)
  Day 20: number analyzed (Participants) | 3 | 2
  Day 20 | 1.33333 (1.15470) | 0 (0)
  Day 21: number analyzed (Participants) | 0 | 2
  Day 21 |  | 0 (0)

3. Secondary Outcome: Pain Score During the Previous 24 Hours
Description: A score ranging from 0 to 10, measured by age appropriate validated pain scale. Because there was only one patient during day 21 time point for this treatment group, the mean and standard deviation could not be calculated.Infants and toddlers (less than age 4 years) or other children who cannot self report, use the FLACC Scale Score each component as a subscore (face, legs, activity, cry, consolability) Total subscores to determine FLACC score Older children (ages 4 to 7 years) who can self-report, use the Faces Pain Scale-Revised (FPS-R) Ages >7 years, Self report using a numeric scale 0-10 without reference to Faces Pain Scale-Revised (FPS-R) Pain score 0 means no pain and 10 means worst pain.The scale information for the FLACC and FPS-R scales are similar.
Time Frame: Daily beginning day 1 through a maximum of 21 days
Population: There were participants in the Gabapentin and Placebo groups that did not have pain assessments at various time points. Pain score was 0 for each placebo participant on days 20 and 21.
Measure: Mean (Standard Deviation); unit: score on a scale 0-10
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 24
score on a scale 0-10
  Day 1 | 3.48000 (2.50200) | 3.41667 (2.39414)
  Day 2 | 3.16000 (2.37487) | 2.20833 (2.14637)
  Day 3 | 3.08000 (2.28983) | 1.87500 (1.87228)
  Day 4 | 2.80000 (2.43242) | 2.12500 (2.64267)
  Day 5 | 2.80000 (2.61406) | 2.00000 (2.14679)
  Day 6 | 2.28000 (1.92614) | 1.91667 (2.20507)
  Day 7 | 2.96000 (2.22636) | 1.16667 (1.60615)
  Day 8: number analyzed (Participants) | 25 | 23
  Day 8 | 2.76000 (2.24128) | 1.69565 (1.91726)
  Day 9: number analyzed (Participants) | 25 | 23
  Day 9 | 2.16000 (2.21133) | 1.34783 (1.74795)
  Day 10: number analyzed (Participants) | 25 | 23
  Day 10 | 2.16000 (2.24870) | 1.43478 (1.64665)
  Day 11: number analyzed (Participants) | 25 | 23
  Day 11 | 2.32000 (2.05589) | 1.56522 (1.67403)
  Day 12: number analyzed (Participants) | 24 | 23
  Day 12 | 2.41667 (2.43018) | 1.52174 (1.90381)
  Day 13: number analyzed (Participants) | 24 | 23
  Day 13 | 2.50000 (2.20671) | 1.60870 (1.85225)
  Day 14: number analyzed (Participants) | 23 | 23
  Day 14 | 2.60870 (2.27115) | 1.56522 (1.64665)
  Day 15: number analyzed (Participants) | 22 | 23
  Day 15 | 2.54545 (2.15423) | 1.39130 (1.67167)
  Day 16: number analyzed (Participants) | 17 | 16
  Day 16 | 2.23529 (1.82104) | 1.56250 (1.82460)
  Day 17: number analyzed (Participants) | 15 | 14
  Day 17 | 1.40000 (1.59463) | 1.92857 (2.01778)
  Day 18: number analyzed (Participants) | 11 | 12
  Day 18 | 2.36364 (3.00908) | 1.00000 (1.65145)
  Day 19: number analyzed (Participants) | 5 | 5
  Day 19 | 1.40000 (1.34164) | 0.40000 (0.89443)
  Day 20: number analyzed (Participants) | 3 | 2
  Day 20 | 2.33333 (0.57735) | 0 (0)
  Day 21: number analyzed (Participants) | 0 | 2
  Day 21 |  | 0 (0)

ADVERSE EVENTS:
Time Frame: through study completion, up to 21 days
Description: Adverse events will be submitted by a member of the study team to the IRB using the existing institutional online reporting mechanisms. All study-related AEs will be collected in the database, regardless of their grade.
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 5/25 | 5/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=25) | Placebo (N=24)
Depressed level of consciousness (Nervous system disorders) | 5 (5) | 5 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT01506453/Prot_SAP_000.pdf